CLINICAL TRIAL: NCT02815488
Title: A Randomised, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of CHF 6297 After Single and Repeated Ascending Doses in Healthy Male Subjects Followed by a Repeated Dose in COPD Patients and a 2-way, Crossover, Double-blind, Placebo-controlled, Repeated Dose Part to Investigate the Anti-inflammatory Effect of CHF 6297 After Lipopolysaccaride (LPS) Challenge in Healthy Male Subjects
Brief Title: A Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Repeat Doses of CHF6297 in Healthy Subjects and Patients With COPD
Acronym: CHF6297 FIH
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Very poor recruitment in the Part 4 of the study
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCD-06297AA1-01; 2015-003075-30 (EudraCT Number)
Record Dates: First submitted 2016-05-25; First posted 2016-06-28 (Estimated); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHF6297 Active (Experimental)
  Interventions: Drug: CHF6297 (Part 1 - SAD); Drug: CHF6297 (Part 2 - MAD); Drug: CHF6297 (Part 3); Drug: CHF6297 (Part 4)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (Part 1 - SAD); Drug: Placebo (Part 2 - MAD); Drug: Placebo (Part 3); Drug: Placebo (Part 4)

INTERVENTIONS:
Drug: CHF6297 (Part 1 - SAD) — Single doses of CHF6297 at each period (for up to 3 periods per subject)
  Arms: CHF6297 Active
Drug: Placebo (Part 1 - SAD) — Single doses of placebo matching CHF6297 at each period (for up to 3 periods per subject)
  Arms: Placebo
Drug: CHF6297 (Part 2 - MAD) — Twice daily doses of CHF6297 for 7 days
  Arms: CHF6297 Active
Drug: Placebo (Part 2 - MAD) — Twice daily doses of placebo matching CHF6297 for 7 days
  Arms: Placebo
Drug: CHF6297 (Part 3) — Twice daily doses of CHF6297 for 14 days
  Arms: CHF6297 Active
Drug: Placebo (Part 3) — Twice daily doses of placebo matching CHF6297 for 14 days
  Arms: Placebo
Drug: CHF6297 (Part 4) — Twice daily doses of CHF6297 for 7 days
  Arms: CHF6297 Active
Drug: Placebo (Part 4) — Twice daily doses of placebo matching CHF6297 for 7 days
  Arms: Placebo

SUMMARY:
CHF6297 is a potent and selective inhibitor of human MAP kinase p38 being developed as an anti-inflammatory agent for the treatment of inflammatory airways diseases. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of single and repeat doses of CHF6297 as dry powder formulation in healthy subjects and in COPD patients. This study is the first administration in humans.

The study will comprise four parts:

Part 1 will consist of two cohorts of healthy male subjects to assess the safety, tolerability and pharmacokinetics of Single Ascending Dose (SAD) of CHF6297.

Part 2 will consist of four cohorts of healthy male subjects to assess the safety, tolerability and pharmacokinetics of Multiple Ascending Dose (MAD) of CHF6297.

Part 3 will consist of one cohort of COPD patients to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of a repeat dose of CHF6297

Part 4 will consist of one cohort of healthy subjects to assess the anti-inflammatory effect of a repeat dose of CHF6297 after LPS challenge.

ELIGIBILITY:
Inclusion criteria:

Part 1, Part 2, Part 4 (Healthy subjects):

* Male subjects aged 18-55 years;
* Non smokers
* Lung function above 80% of predicted normal value
* Healthy subjects based on medical evaluation including medical history, physical examination, laboratory tests and cardiac testing
* ability to produce an adequate induced sputum sample (study part 4 only)

Part 3 (COPD patients):

* Males and females aged 40-75 years
* Current or past smokers
* stable patients with a post-bronchodilator FEV1 between 40 and 80% of predicted normal value and FEV1/FVC ratio <0.7
* Ability to produce a spontaneous and an adequate induced sputum sample

Exclusion Criteria:

Parts 1,2, 4 (Healthy subjects):

* Any clinically relevant abnormalities and/or uncontrolled diseases
* Abnormal laboratory values
* Recent respiratory tract infection
* Hypersensitivity to the drug or excipients
* Positive serology results
* Positive cotinine, alcohol, drug of abuse tests

Part 3 (COPD patients):

* Females of childbearing potential
* History of asthma
* Unstable concomitant diseases
* Abnormal relevant Holter ECG parameters
* Recent acute exacerbations of COPD or respiratory tract infection
* Hypersensitivity to the drug or excipients
* Positive serology results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Adverse events | Part 1 from Day 1 until Day 4, Part 2 from Day 1 until Day 8, Part 3 from Day 1 until Day 17, Part 4 from Day 1 until Day 8
  Treatment-related Adverse events
Change in Vital signs | Part 1 from Day 1 until Day 4, Part 2 from Day 1 until Day 8, Part 3 from Day 1 until Day 17
  Blood pressure
Change in Holter ECG parameters | Part 1 Day 1-2, Part 2 Day 1-2 and Day 7-8, Part 3 Day 1-2 and Day 14-15
  HR, QTcF, PR, QRS + holter recording abnormalities
Change in FEV1 | Part 1 Day 1-2, Part 2 Day 1 and Day 7-8, Part 3 Day 1, Day 10 and Day 14
  Forced exhalation volume in the first second
Change in Laboratory parameters | Part 1 Day 1 and Day 4, Part 2 Day 1 and Day 8, Part 3 Day 1 and Day 15
  Clinical chemistry and haematology + urinalysis

SECONDARY OUTCOMES:
Area under the plasma concentration vs time curve | Part 1 Day 1 until Day 4, Part 2 Day 1 and Day 7, Part 3 Day 1 and Day 14
Peak plasma concentration (Cmax) | Part 1 Day 1 until Day 4, Part 2 Day 1 and Day 7, Part 3 Day 1 and Day 14
  maximum plasma concentration of CHF6297
Time to reach the maximum plasma concentration (tmax) | Part 1 Day 1 until Day 4, Part 2 Day 1 and Day 7, Part 3 Day 1 and Day 14
Elimination half-life (t1/2) | Part 1 Day 1 until Day 4, Part 2 Day 1 and Day 7, Part 3 Day 1 and Day 14
Clearance (CL/F) | Part 1 Day 1 until Day 4, Part 2 Day 1 and Day 7, Part 3 Day 1 and Day 14
  Absolute plasma clearance
Volume of distribution (Vz/F) | Part 1 Day 1 until Day 4, Part 2 Day 1 and Day 7, Part 3 Day 1 and Day 14
  plasma volume of distribution
Urinary excretion (Ae) | Part 1 from Day 1 to Day 4, Part 2 Day 1 and Day 7
  Amount of CHF6297 excreted in urine
fraction excreted (fe) | Part 1 from Day 1 to Day 4, Part 2 Day 1 and Day 7
  Percentage of drug excreted in urine
Renal clearance (CLr) | Part 1 from Day 1 to Day 4, Part 2 Day 1 and Day 7

OTHER OUTCOMES:
Part 3: markers of inflammation (exploratory) | after 14 days of dosing
  Blood and sputum biomarkers
Part 4: markers of inflammation (exploratory) | after 7 days of dosing
  Blood and sputum biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MD, Principal Investigator — Quotient Clinical; Dave Singh, MD, Principal Investigator — Medicines Evaluation Unit
Locations (2):
- United Kingdom (2):
  - Quotient Clinical, Ruddington, Nottingham
  - Medicines Evaluation Unit, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2015-003075-30/results